CLINICAL TRIAL: NCT06231615
Title: Efficacy of Fascia Exercises in Migraine Patients: A Randomized Controlled Trial
Brief Title: Efficacy of Fascia Exercises in Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07.04.2022/06
Record Dates: First submitted 2024-01-03; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Migraine
Keywords: migraine; pain; exercise; fascia
MeSH Terms: conditions — Migraine Disorders; Pain; Motor Activity | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: dual parallel group design
Who Masked: Outcomes Assessor
Masking Description: The evaluation of the patients was carried out by a blinded investigator, and the treatment was carried out by a different investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients in this group are the group to which fascia exercises are applied.
  Interventions: Other: Fascia exercises; Other: Conventional physiotherapy and breathing exercises
- Control group (Other): Patients in this group are the group to which conventional physiotherapy and breathing exercises are applied.
  Interventions: Other: Conventional physiotherapy and breathing exercises

INTERVENTIONS:
Other: Fascia exercises — Fascia exercises are slow and calm movements similar to yoga performed by the person herself/himself.
  Arms: Treatment group
Other: Conventional physiotherapy and breathing exercises — Head and neck exercises and breathing exercises

SUMMARY:
Migraine, which is characterized by attacks and many accompanying symptoms, negatively affects the quality of life of patients. Although different methods have been tried for migraine, there is no definitive treatment approach yet. The aim of this study is to examine the effect of fascia exercises as a new approach on the symptoms and complaints of migraine patients.

The study was completed with 30 volunteer migraine patients. Participants were divided into two groups in a randomized controlled manner. While head-neck and breathing exercises were applied to the control group, fascial pattern exercises were performed in the study group in addition to these exercises. This protocol was applied 2 days a week for 6 weeks. Pain intensity, quality of life and sleep, heart rate changes, depression and anxiety levels and satisfaction levels were evaluated before and after the treatment.

Fascial pattern exercises are an effective approach on the symptoms and complaints of migraine patients and can be adopted as a complementary application in migraine treatment. Since this is the first study in this field, it needs to be supported by other studies in order to increase the provability of the effectiveness of the exercises.

DETAILED DESCRIPTION:
Migraine, which is characterized by attacks and many accompanying symptoms, negatively affects the quality of life of patients. Although different methods have been tried for migraine, there is no definitive treatment approach yet. The aim of this study is to examine the effect of fascia exercises as a new approach on the symptoms and complaints of migraine patients.

The study was completed with 30 volunteer migraine patients. Participants were divided into two groups in a randomized controlled manner. While head-neck and breathing exercises were applied to the control group, fascial pattern exercises were performed in the study group in addition to these exercises. This protocol was applied 2 days a week for 6 weeks. Pain intensity, quality of life and sleep, heart rate changes, depression and anxiety levels and satisfaction levels were evaluated before and after the treatment.

Demographic and descriptive characteristics of the participants were similar (p>0.05). In both groups, the number of attacks, duration of attacks, pain intensity, migraine-related disability and anxiety levels decreased and sleep quality improved after treatment (p<0.05). There was no significant difference in heart rate change parameters within and between the groups (p>0.05). There was no significant difference between the groups in terms of treatment efficacy (p>0.05). Patient satisfaction was higher in the fascia exercises group (p<0.05).

Fascial pattern exercises are an effective approach on the symptoms and complaints of migraine patients and can be adopted as a complementary application in migraine treatment. Since this is the first study in this field, it needs to be supported by other studies in order to increase the provability of the effectiveness of the exercises.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis of migraine for at least one year
* between the ages of 18-65 years,
* having migraine attacks at least 5 days a month,
* having a history of migraine starting under the age of 50,
* giving informed written consent to participate in the study

Exclusion Criteria:

* headache due to organic or secondary causes (history of subarachnoid or cerebral hemorrhage, hypertension, cerebral embolism or thrombosis),
* receiving acupuncture treatment in the last 6 months,
* history of bleeding diathesis or receiving anticoagulant treatment,
* being pregnant or lactating,
* history of malignancy,
* having a diagnosis of depression or receiving antidepressant treatment,
* caffeine consumption in the last 4 hours,
* tobacco use in the last 48 hours,
* drug and alcohol use in the last week,
* eating within 2 hours prior to the test,
* being unable to move independently,
* having an uncontrolled medical condition,
* chronic cardiovascular disease,
* recent surgery,
* symptoms of somatic dysfunction,
* musculoskeletal injuries,
* any medication that interferes with the autonomic nervous system or immune system (e.g., beta blockers, steroids, or TNF-a inhibitors)
* any medical condition that affects the autonomic nervous system or immune system

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | Change from baseline at 6 weeks treatment program
  Heart rate variability is a tool that allows the investigation of cardiovascular autonomic function through the measurement of variations in RR intervals and provides valuable information about the control of the autonomic nervous system

SECONDARY OUTCOMES:
Pain level | Change from baseline at 6 weeks treatment program
  Visual analog scale was used to examine pain levels of participants.Individuals are presented with a line numbered evenly from 1 to 10 and asked to mark the point corresponding to their pain intensity. A higher score indicates that the severity of pain is increasing.
Level of disability due to migraine | Change from baseline at 6 weeks treatment program
  The Migraine Disability Scale was used to evaluate the level of disability due to headache.Patients answer the questions by reflecting on their last 3 months. The total score is examined in 4 stages. 0-5 points means stage 1, 6-10 points means stage 2, 11-20 points means stage 3, 21 points and above means stage 4. 21 points and above means serious disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be available to the responsible researcher.